CLINICAL TRIAL: NCT02264886
Title: Pilot Study of Online, Adaptive MRI-Guided SBRT for Unresectable Primary or Oligometastatic Central Thorax and Abdominal Malignancies
Brief Title: Adaptive MRI-Guided SBRT for Unresectable Primary or Oligometastatic Central Thorax and Abdominal Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201410002
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Central Thorax Cancer; Liver Cancer; Non-Liver Abdominal Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: Stereotactic body radiation therapy (Experimental): Radiotherapy will consist of stereotactic body therapy, to be given over five fractions, delivered once daily or once every other day for a period of one to two weeks, for a total of five treatments.
  All patients will undergo MRI simulation in positioning appropriate for the specific treatment site. When medically feasible and applicable, patients will be simulated with IV and small bowel contrast (for non-thorax cases).
  Interventions: Radiation: MRI-guided stereotactive body radiation therapy

INTERVENTIONS:
Radiation: MRI-guided stereotactive body radiation therapy
  Other Names: SBRT

SUMMARY:
The purpose of this research study is evaluate whether it's feasible to give radiation therapy using an MRI-guided adaptive technique. MRI-guided adaptive radiation therapy involves the adjustment or re-planning of treatment day by day while the participant is receiving treatment. The adaptive technique has previously been used in a different fashion to adjust the treatment plan after the fact, but using MRI scanning to re-plan treatment while the participant is still on the table is a new way of using the adaptive technique. This may allow doctors to use more radiation to treat the tumor while better protecting normal tissues. A special radiation treatment machine incorporates both an MRI scanner and radiation treatment devices so that the planning and treatment can be done using the same machine.

DETAILED DESCRIPTION:
In this trial, the feasibility of delivering online, adaptive MRI-guided stereotactic body radiation therapy for oligometastatic disease using a novel, integrated Co-60-MRI machine will be evaluated. To best assess this technology, we will focus on three specific oligometastatic disease sites that have historically highlighted the limitations of SBRT. Specifically, we will enroll patients with oligometastatic disease of the central thorax, liver, and non-liver abdomen to receive adaptive, MRI-guided SBRT with MRI simulation and MRI treatment gating. Patients will be treated in five fractions over one to two weeks. By adhering to strict normal tissue constraints, expected toxicity will be within the current standard of care, but allow adaptation based on daily anatomic changes. The prescription dose will be determined based on above hard normal tissue constraints, and capped at 15 Gy per fraction. Although our long-term goal will be to achieve improved local control and disease-free survival with reduced toxicity, the present study will be driven by short-term goals of demonstrating feasibility of an on-table adaptive approach, which has never previously been reported.

ELIGIBILITY:
Inclusion Criteria:

* Oligometastatic or unresectable primary disease planned for SBRT with biopsy-proven primary disease histology of solid tumor categorization with the exception of small cell cancers.
* Must be deemed medically fit for SBRT to the liver or lung by the treating physician.
* At least 18 years of age.
* Karnofsky performance status > 60 (see Appendix A)
* Must have completed any systemic therapy at least one week prior to planned start of SBRT (two weeks preferred), and must have no plans to initiate systemic therapy for at least one week following end of SBRT (two weeks preferred).
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Primary disease of hematologic origin, lymphoma, or small cell cancer.
* Past history of radiotherapy within the projected treatment field of any of the disease sites to be treated by MRI-guided, online adaptive SBRT.
* Widespread progressive disease, i.e., more than 3 sites of progressive disease (more than 3 sites of disease are permitted provided there are no more than 3 sites of progressive disease).
* Currently receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of study entry.
* Medical contraindication to undergoing MR imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of the online, adaptive, MRI-guided SBRT | Average time of 2 weeks
  Feasibility is determined that confirming that the treatment can be delivered with less than 80 minutes total treatment (on table) time, for more than 75% of cases where treatment adaptation is indicated.

SECONDARY OUTCOMES:
Tumor response rate | 3 months
Local, in-field control rate | 6 months
Progression free survival rate (PFS) | 6 months
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Disease free survival rate | 6 months
Overall survival rate | 6 months
Patient-reported quality of life | 6 months
  Using the EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Parag J Parikh, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu